CLINICAL TRIAL: NCT02674087
Title: Prospective Monitoring of Children Born in Haute Vienne From Uterine Life to Adulthood
Acronym: NEHAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Collaborators: Fondation Patrtenariale Unilim (Unknown); ARS (Unknown); La poste (Unknown)
Responsible Party: Sponsor
Other Study IDs: I1 029
Record Dates: First submitted 2014-04-14; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Child Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Expectant women

SUMMARY:
The purpose of this survey is to collect data from intrauterine life until the age of 18 of children born in Haute Vienne.

The interest to realize such survey is to find correlations and interactions that may exist between the events that occurred during intrauterine life and those that will occur after the birth of the child. The investigators will examine every aspect of these children's lives from the perspectives of health, social sciences and environmental health

These are medical events (occurrence of disease, medication), but also socio-cultural for this child (living environment, exposure to possible contaminants, events in family history).

This cohort aims to include 3000 children a year (whose parents consented to their inclusion), all born at Haute-Vienne.

ELIGIBILITY:
Inclusion Criteria:

* Any child born in one of the three maternity hospitals in the Haute-Vienne (CHU Limoges, Clinique des Emailleurs, Hospital Saint-Junien).
* Any child who's parents consented to their inclusion.

Exclusion Criteria:

* Children born at home.
* Children abandoned at birth.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Expectant mother
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Rate of enrollment | At 3 years
  3 years after the study has started, the investigators will evaluate the rate of enrollment.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Clinique des Emailleurs, Limoges
  - HME, Limoges
  - Centre Hositalier de Saint Junien, Saint-Junien